CLINICAL TRIAL: NCT01134315
Title: A Prospective, Multicenter Study to Evaluate the Safety of Paricalcitol Capsules as Determined by Hypercalcemia in Pediatric Patients Ages 0 to 16 With Chronic Kidney Disease (CKD) Stage 5 Receiving Peritoneal Dialysis (PD) Within Current Clinical Practice
Brief Title: Study to Evaluate Safety of Vitamin D Receptor Activators in Patients Ages 0 to 16 With Chronic Kidney Disease Stage 5 Receiving Peritoneal Dialysis Within Current Clinical Practice
Status: Terminated | Type: Observational
Why Stopped: Terminated after FDA agreement.
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: North America Pediatric Renal Trials and Collaborative Studies (NAPRTCS) (Unknown)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-053
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Results first posted 2013-08-13 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-05

CONDITIONS: Secondary Hyperparathyroidism; End-Stage Renal Disease
Keywords: Evaluating incidence of hypercalcemia in pediatric patients
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Kidney Failure, Chronic | interventions — paricalcitol; Calcitriol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Paricalcitol: Pediatric participants who received paricalcitol capsules to treat secondary hyperparathyroidism (SHPT). Paricalcitol was prescribed by each physician under the usual and customary practice of that physician.
  Interventions: Drug: Paricalcitol
- Calcitriol: Pediatric participants who received calcitriol to treat secondary hyperparathyroidism (SHPT). Calcitriol was prescribed by each physician under the usual and customary practice of that physician.
  Interventions: Drug: Calcitriol

INTERVENTIONS:
Drug: Paricalcitol
  Other Names: ABT-358; Zemplar
  Groups: Paricalcitol
Drug: Calcitriol
  Groups: Calcitriol

SUMMARY:
The objective of this study was to observe the safety of paricalcitol utilization in pediatric participants (ages 0 to 16 years old) being treated for secondary hyperparathyroidism (SHPT). Participants were to be followed for a minimum of 3 months and up to approximately 36 months to monitor the incidence of hypercalcemia (high calcium levels in blood).

DETAILED DESCRIPTION:
Investigators were free to determine the appropriate therapy for each participant based on clinical judgment. Decisions to prescribe paricalcitol or calcitriol were made independently prior to enrollment of participants in this observational study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 0 to 16 years of age (inclusive), on peritoneal dialysis for at least 30 days.
2. The patient has a history of secondary hyperparathyroidism as defined by having initiated a vitamin D receptor activator to treat an elevated parathyroid hormone level.
3. The patient is attending a site associated with North America Pediatric Renal Trials and Collaborative Studies (NAPRTCS) Dialysis Registry.
4. Patient and the patient's parent or legal guardian must voluntarily sign and date an informed consent and/or assent, approved by the local Independent Ethics Committee/Institutional Review Board, prior to the initiation of any screening or study-specific procedures.
5. Patient has received paricalcitol or calcitriol for a minimum of 10 days.

Exclusion Criteria:

1. Patient is scheduled for a kidney transplant within 3 months.
2. Patient is expected to stop peritoneal dialysis within 3 months.
3. Patient is expected to transfer to hemodialysis within 3 months.
4. Patient is planning to be enrolled in an investigational study where the drug and/or dose are unknown to the investigator within the first 3 months from the date of patient enrollment.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This was a multicenter, United States only study of pediatric (0 to 16 years) males and females receiving peritoneal dialysis, treated in a routine clinical setting. Patients were recruited from private nephrology practices or hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2010-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Eldred, MD, Study Director — AbbVie
Locations (18):
- United States (18):
  - Site Reference ID/Investigator# 37082, Birmingham, Alabama
  - Site Reference ID/Investigator# 26762, Gainesville, Florida
  - Site Reference ID/Investigator# 28529, Orlando, Florida
  - Site Reference ID/Investigator# 26748, Atlanta, Georgia
  - Site Reference ID/Investigator# 37582, New Orleans, Louisiana
  - Site Reference ID/Investigator# 39973, Baltimore, Maryland
  - Site Reference ID/Investigator# 26769, Boston, Massachusetts
  - Site Reference ID/Investigator# 26768, Detroit, Michigan
  - Site Reference ID/Investigator# 26747, Kansas City, Missouri
  - Site Reference ID/Investigator# 26749, Akron, Ohio
  - Site Reference ID/Investigator# 26751, Cincinnati, Ohio
  - Site Reference ID/Investigator# 26765, Columbus, Ohio
  - Site Reference ID/Investigator# 28528, Oklahoma City, Oklahoma
  - Site Reference ID/Investigator# 26763, Portland, Oregon
  - Site Reference ID/Investigator# 28526, Charlottesville, Virginia
  - Site Reference ID/Investigator# 26758, Seattle, Washington
  - Site Reference ID/Investigator# 40382, Madison, Wisconsin
  - Site Reference ID/Investigator# 26759, Wauwatosa, Wisconsin

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paricalcitol | Calcitriol
Started | 21 | 40
Completed | 12 (Completed study drug treatment during the observational study (ie, prior to study termination).) | 21 (Completed study drug treatment during the observational study (ie, prior to study termination).)
Not Completed | 9 | 19
Not completed — Adverse Event | 1 | 2
Not completed — Other Reason | 8 | 17

BASELINE CHARACTERISTICS:
Groups:
- Paricalcitol: Pediatric participants who received paricalcitol capsules to treat SHPT. Paricalcitol was prescribed by each physician under the usual and customary practice of that physician.
- Calcitriol: Pediatric participants who received calcitriol to treat SHPT. Calcitriol was prescribed by each physician under the usual and customary practice of that physician.
- Total: Total of all reporting groups
Arm/Group | Paricalcitol | Calcitriol | Total
Number analyzed (Participants) | 21 | 40 | 61
Age, Customized [Number; unit: participants]
  <8 years | 5 | 19 | 24
  >=8 years | 16 | 21 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 19
  Male | 14 | 28 | 42
Region of Enrollment [Number; unit: participants]
  United States | 21 | 40 | 61

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Incidence of Hypercalcemia
Description: Hypercalcemia was defined as calcium >10.2 mg/dL. Percentage of participants with hypercalcemia is presented for the overall population, the subgroup of participants in the study for less than 3 months, and those in the study for greater than or equal to 3 months.
Time Frame: Monitored from time of informed consent through end of study + 30 days (total of 745 days).
Population: All Treated Population (all participants who received at least 1 dose of paricalcitol [paricalcitol group] or at least one dose of calcitriol [calcitriol group]).
Measure: Number; unit: percentage of participants
Arm/Group | Paricalcitol | Calcitriol
Number analyzed (Participants) | 19 | 37
percentage of participants
  Overall population (n=19, 37) | 36.8 | 54.1
  Participants <3 months in study (n=2, 5) | 50.0 | 0
  Participants >=3 months in study (n=17, 32) | 35.3 | 62.5

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs), Serious AEs (SAEs), Deaths and Discontinuations Due to AEs
Description: AE: any untoward medical occurrence that does not necessarily have a causal relationship with treatment; any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered causally related to the use of the product (either paricalcitol or calcitriol); can result from use of the drug as stipulated in the labeling, as well as from accidental or intentional overdose, drug abuse, or drug withdrawal; any worsening of a pre-existing condition or illness. Severity was categorized as mild, moderate, or severe. SAE: AE that results in the death; is life-threatening; results in hospitalization or prolongation of hospitalization; is a congenital anomaly; results in persistent or significant disability/incapacity; is an important medical event requiring medical or surgical intervention to prevent serious outcome; is a spontaneous or elective abortion. For more details, please see the AE section of this record.
Time Frame: Monitored from time of informed consent through end of study + 30 days (total of 745 days).
Population: All participants
Measure: Number; unit: participants
Arm/Group | Paricalcitol | Calcitriol
Number analyzed (Participants) | 21 | 40
participants
  Any AE | 17 | 32
  Any severe AE | 3 | 12
  Any SAE | 8 | 26
  Any AE leading to discontinuation of study drug | 1 | 3
  Any AE leading to discontinuation of study | 0 | 1
  Any fatal AE | 0 | 2
  Deaths (includes non-treatment-emergent deaths) | 0 | 2

3. Secondary Outcome: Mean Baseline (BL) and Change From Baseline in Potassium, Sodium, Chloride, Bicarbonate at Final Visit (FV)
Description: Normal ranges for these chemistry measurements varied according to the age of the participant.
Time Frame: Baseline, Final Visit (defined as the last post-baseline observation, up to end of study [715 days])
Population: All Treated Population (all participants who received at least 1 dose of paricalcitol [paricalcitol group] or at least one dose of calcitriol [calcitriol group]); n=number of participants with measurements at baseline and given time point.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Paricalcitol | Calcitriol
Number analyzed (Participants) | 19 | 37
mEq/L
  Potassium, BL (n=15, 29) | 4.4 (0.70) | 4.4 (0.83)
  Potassium, change from BL at FV (n=15, 29) | -0.1 (0.81) | -0.5 (1.00)
  Sodium, BL (n=15, 29) | 138.0 (2.75) | 139.3 (4.42)
  Sodium, change from BL at FV (n=15, 29) | 0.2 (2.96) | -0.7 (3.43)
  Chloride, BL (n=15, 29) | 99.5 (4.75) | 98.6 (3.78)
  Chloride, change from BL at FV (n=15, 29) | -0.5 (4.52) | -1.1 (4.07)
  Bicarbonate, BL (n=15, 28) | 26.1 (2.76) | 25.9 (4.12)
  Bicarbonate, change from BL at FV (n=15, 28) | 0.2 (3.63) | 0.1 (4.26)

4. Secondary Outcome: Mean Baseline (BL) and Change From Baseline in Calcium, Inorganic Phosphate (IP), Blood Urea Nitrogen (BUN), Creatinine at Final Visit (FV)
Description: Normal ranges for these chemistry measurements varied according to the age of the participant.
Time Frame: Baseline, Final Visit (defined as the last post-baseline observation, up to end of study [715 days])
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Paricalcitol | Calcitriol
Number analyzed (Participants) | 19 | 37
mg/dL
  Calcium, BL (n=15, 30) | 9.2 (0.84) | 9.3 (1.10)
  Calcium, change from BL at FV (n=15, 30) | 0.0 (0.77) | 0.5 (1.22)
  Inorganic Phosphate (IP), BL (n=13, 29) | 5.8 (1.74) | 5.9 (1.71)
  IP, change from BL at FV (n=13, 29) | -0.4 (1.55) | 0.4 (1.89)
  BUN, BL (n=15, 29) | 52.7 (24.43) | 49.8 (18.69)
  BUN, change from BL at FV (n=15, 29) | -10.7 (23.18) | -1.9 (19.05)
  Creatinine, BL (n=15, 29) | 9.4 (4.35) | 8.8 (4.35)
  Creatinine, change from BL at FV (n=15, 29) | 0.3 (1.98) | 0.3 (2.19)

5. Secondary Outcome: Mean Baseline and Change From Baseline in 25-Hydroxy Vitamin D3 at Final Visit (FV)
Description: Normal ranges for these chemistry measurements varied according to the age of the participant.
Time Frame: Baseline, Final Visit (defined as the last post-baseline observation, up to end of study [715 days])
Population: All Treated Population (all participants who received at least 1 dose of paricalcitol [paricalcitol group] or at least one dose of calcitriol [calcitriol group]) with measurements at baseline and given time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Paricalcitol | Calcitriol
Number analyzed (Participants) | 0 | 2
ng/mL
  Baseline |  | 28.4 (6.51)
  Change from Baseline at FV |  | 7.5 (0.78)

6. Secondary Outcome: Mean Baseline and Change From Baseline in 1,25-Dihydroxy Vitamin D3 at Final Visit (FV)
Description: Normal ranges for these chemistry measurements varied according to the age of the participant.
Time Frame: Baseline, Final Visit (defined as the last post-baseline observation, up to end of study [715 days])
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Paricalcitol | Calcitriol
Number analyzed (Participants) | 1 | 0
pg/mL
  Baseline | 20.0 (NA) — Only 1 participant analyzed. |
  Change from Baseline at FV | -10.0 (NA) — Only 1 participant analyzed. |

7. Secondary Outcome: Mean Baseline and Change From Baseline in Parathyroid Hormone at Final Visit (FV)
Description: Normal ranges for these chemistry measurements varied according to the age of the participant.
Time Frame: Baseline, Final Visit (defined as the last post-baseline observation, up to end of study [715 days])
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Paricalcitol | Calcitriol
Number analyzed (Participants) | 15 | 21
pg/mL
  Baseline | 571.7 (532.52) | 592.8 (619.72)
  Change from Baseline at FV | -102.5 (695.39) | -193.4 (489.11)

8. Secondary Outcome: Mean Baseline and Change From Baseline in Albumin at Final Visit (FV)
Description: Normal ranges for these chemistry measurements varied according to the age of the participant.
Time Frame: Baseline, Final Visit (defined as the last post-baseline observation, up to end of study [715 days])
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Paricalcitol | Calcitriol
Number analyzed (Participants) | 15 | 29
g/dL
  Baseline | 3.3 (0.77) | 3.8 (0.52)
  Change from Baseline at FV | -0.0 (0.54) | -0.1 (0.69)

ADVERSE EVENTS:
Time Frame: Monitored from time of informed consent through end of study + 30 days (total of 745 days).
Description: Treatment-emergent events are presented.
Arm/Group | Paricalcitol | Calcitriol
Serious Adverse Events (participants affected / at risk) | 8/21 | 26/40
Other Adverse Events (participants affected / at risk) | 15/21 | 29/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol (N=21) | Calcitriol (N=40)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Middle Ear Effusion (Ear and labyrinth disorders) | 0 | 1
Adrenocortical Insufficiency Acute (Endocrine disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Umbilical Hernia (Gastrointestinal disorders) | 0 | 1
Umbilical Hernia, Obstructive (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Catheter Site Erosion (General disorders) | 1 | 1
Device Dislocation (General disorders) | 0 | 1
Device Leakage (General disorders) | 0 | 1
Device Malfunction (General disorders) | 0 | 1
Medical Device Complication (General disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 3
Bronchiolitis (Infections and infestations) | 0 | 1
Catheter Site Cellulitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1
Device Related Infection (Infections and infestations) | 0 | 1
Fungal Peritonitis (Infections and infestations) | 0 | 1
Meningitis Aseptic (Infections and infestations) | 0 | 1
Otitis Media (Infections and infestations) | 0 | 2
Peritonitis (Infections and infestations) | 4 | 8
Peritonitis Bacterial (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Pneumonia Primary Atypical (Infections and infestations) | 0 | 1
Pseudomonas Infection (Infections and infestations) | 0 | 1
Respiratory Syncytial Virus Bronchiolitis (Infections and infestations) | 0 | 1
Respiratory Tract Infection Viral (Infections and infestations) | 0 | 1
Septic Shock (Infections and infestations) | 1 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Viral Infection (Infections and infestations) | 0 | 1
Peritoneal Dialysis Complication (Injury, poisoning and procedural complications) | 0 | 1
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 1 | 0
Blood Urea Nitrogen/Creatinine Ratio Increased (Investigations) | 0 | 1
Weight Decreased (Investigations) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Failure To Thrive (Metabolism and nutrition disorders) | 0 | 1
Fluid Overload (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Renal Osteodystrophy (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebral Infarction (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 2 | 0
Hypertensive Encephalopathy (Nervous system disorders) | 1 | 0
Seizure Anoxic (Nervous system disorders) | 0 | 1
Eating Disorder (Psychiatric disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 2
Hypertensive Emergency (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Wegener's Granulomatosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol (N=21) | Calcitriol (N=40)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Deafness Neurosensory (Ear and labyrinth disorders) | 1 | 0
Middle Ear Effusion (Ear and labyrinth disorders) | 0 | 1
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 0 | 1
Visual Impairment (Eye disorders) | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 1
Abdominal Mass (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 4
Bloody Peritoneal Effluent (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 5
Gastritis (Gastrointestinal disorders) | 1 | 0
Impaired Gastric Emptying (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1
Lip Swelling (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 5
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Retching (Gastrointestinal disorders) | 0 | 2
Umbilical Hernia (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 4
Asthenia (General disorders) | 1 | 0
Catheter Site Discharge (General disorders) | 0 | 1
Catheter Site Erythema (General disorders) | 0 | 2
Catheter Site Haemorrhage (General disorders) | 0 | 1
Catheter Site Pain (General disorders) | 0 | 1
Catheter Site Related Reaction (General disorders) | 0 | 1
Device Damage (General disorders) | 0 | 1
Device Malfunction (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 2
Oedema Peripheral (General disorders) | 1 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 4
Seasonal Allergy (Immune system disorders) | 1 | 0
Candida Nappy Rash (Infections and infestations) | 0 | 1
Catheter Site Infection (Infections and infestations) | 2 | 3
Cellulitis (Infections and infestations) | 2 | 0
Chronic Sinusitis (Infections and infestations) | 1 | 0
Clostridial Infection (Infections and infestations) | 0 | 1
Conjunctivitis Infective (Infections and infestations) | 0 | 1
Device Related Infection (Infections and infestations) | 2 | 1
Ear Infection (Infections and infestations) | 1 | 3
Eye Infection (Infections and infestations) | 0 | 1
Fungal Infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Graft Infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Oral Herpes (Infections and infestations) | 0 | 1
Otitis Media (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 2 | 3
Pharyngitis Streptococcal (Infections and infestations) | 3 | 2
Pneumonia (Infections and infestations) | 0 | 1
Pseudomonas Infection (Infections and infestations) | 0 | 1
Respiratory Tract Infection Viral (Infections and infestations) | 0 | 2
Serratia Infection (Infections and infestations) | 0 | 1
Staphylococcal Infection (Infections and infestations) | 0 | 1
Stitch Abscess (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 5
Wound Infection (Infections and infestations) | 2 | 0
Arteriovenous Fistula Site Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Feeding Tube Complication (Injury, poisoning and procedural complications) | 0 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Blood Cortisol Increased (Investigations) | 1 | 0
Blood Glucose Increased (Investigations) | 0 | 1
Blood Parathyroid Hormone Increased (Investigations) | 1 | 0
Blood Phosphorus Decreased (Investigations) | 0 | 1
Blood Phosphorus Increased (Investigations) | 1 | 0
Blood Pressure Increased (Investigations) | 0 | 1
Haemoglobin Decreased (Investigations) | 1 | 0
Heart Rate Increased (Investigations) | 0 | 1
Occult Blood Positive (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal Osteodystrophy (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebral Haemorrhage (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 2
Lethargy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Listless (Psychiatric disorders) | 0 | 1
Menstrual Disorder (Reproductive system and breast disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Increased Viscosity Of Bronchial Secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling Face (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 3
Hypotension (Vascular disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.